CLINICAL TRIAL: NCT03166384
Title: A Prospective Randomized Study Comparing Surgery Using Electrosurgical Bipolar Sealing Devices and Surgery Using Conventional Electro-cautery
Brief Title: ELectrosurgical Bipolar Devices VS Conventional Electro-cauterization in Breast Surgery
Acronym: ELBCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Hyung Seok Park, MD, PhD, Clinical Assistant Professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-2017-0002
Record Dates: First submitted 2017-05-21; First posted 2017-05-25 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Seroma as Procedural Complication
Keywords: electrosurgical bipolar sealing devices, breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- control group (Active Comparator): For the patients in the control group, surgeon dose not use electrosurgical bipolar sealing device at all and use conventional tie and ligation methods during tissue dissection and vessel ligation.
  interventions: 'conventional suture and tie'
  Interventions: Procedure: conventional suture and tie
- study group (Experimental): For the patients in the study group, the surgeon uses electrosurgical bipolar sealing device during tissue dissection and vessel ligation as much as possible.
  interventions: electrosurgical bipolar sealing devices
  Interventions: Device: electrosurgical bipolar sealing devices

INTERVENTIONS:
Device: electrosurgical bipolar sealing devices — Electrosurgical bipolar sealing devices use the body's own collagen and elastin to create a permanent fusion zone through a combination of pressure and energy. Previous studies suggested that surgery using these devices lead to significant decrease of seroma formation, however their advantages are not well established in case of mastectomy for breast cancer.
  Arms: study group
Procedure: conventional suture and tie — the surgeon uses electrosurgical bipolar sealing device during tissue dissection and vessel ligation as much as possible.
  Arms: control group

SUMMARY:
There was no study about application of electrosurgical bipolar sealing device for mastectomy in Korean population, because Korean national insurance did not cover use of the advanced sealing device until last year. Sample size of the previous studies was too small to draw a solid conclusion. Therefore, this study was designed prospectively to evaluate whether application of bipolar energy device for mastectomy could provide clinical benefit in terms of reducing seroma formation.

DETAILED DESCRIPTION:
Lymphorrhea and seroma are the most common complications of mastectomy in patients with breast cancer. Seroma formation increases admission period, follow-up duration, and postoperative discomforts. Repeated aspiration of seroma increases risk of re-admission due to wound infection. Seroma formation after mastectomy occurs in 10% to 85% of cases with mastectomy. Known risk factors according to previous studies are old age(>60 years), high BMI, tumor size, preoperative chemotherapy, surgical extent, and number of retrieved lymph nodes. To reduce postoperative complications including seroma formation, meticulous hemostasis and lymphatic ligation technique are necessary.

Procedures using new surgical devices such as bipolar sealing devices have been introduced. Electrosurgical bipolar sealing devices use the body's own collagen and elastin to create a permanent fusion zone through a combination of pressure and energy. Previous studies suggested that surgery using these devices lead to significant decrease of seroma formation, however their advantages are not well established in case of mastectomy for breast cancer. Several studies showed that an advanced sealing system like bipolar energy sealing system can reduce operative time and cost for postoperative management compared to conventional clamp and tie method in non-breast surgery.

If electrosurgical bipolar sealing devices are applied during mastectomy, there would be several potential benefits on vessel and lymphatic ligation. Conventional ligation and monopolar cauterization have several weak points including incompletion of ligation and thermal injury during procedures. On the other hand, electrosurgical bipolar sealing devices can provide a combination of pressure and energy simultaneously to minimize thermal injury and create a permanent fusion zone.

Previous studies suggested that electrosurgical bipolar sealing devices shortened removal time of drain after axillary lymph node dissection compared with conventional methods. Another study reported benefits on reducing blood loss, drainage amount, and length of hospital stay. Moreover, a recent study also reported that skin sparing mastectomy using electrosurgical bipolar sealing devices can be used in patients with breast cancer.

However, there are several limitations in previous studies. There was no study about application of electrosurgical bipolar sealing device for mastectomy in Korean population, because Korean national insurance did not cover use of the advanced sealing device until last year. Sample size of the previous studies was too small to draw a solid conclusion. Therefore, this study was designed prospectively to evaluate whether application of bipolar energy device for mastectomy could provide clinical benefit in terms of reducing seroma formation.

ELIGIBILITY:
Inclusion Criteria:

* 20 years old and over
* Patients planned to undergo total mastectomy and axillary lymph node dissection
* Patients planned to undergo total mastectomy and sentinel lymph node biopsy and/or reconstruction
* Patients planned to undergo partial mastectomy and axillary lymph node dissection

Exclusion Criteria:

* Bilateral breast cancer patients
* Male breast cancer patients
* Patients who underwent ipsilateral axillar surgery or axillar radiation therapy
* Recurrent breast cancer patients
* Patients who cannot give informed consents such as non-Korean speakers and patients with intellectual disabilities
* Vulnerable patients such as pregnant women for enrollment
* Patients without drain catheter
* Patients with Ductal carcinoma in situ who have not undergone ipsilateral sentinel lymph node biopsy or axillar lymph node dissection

Ages: 20 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Total drainage volume after surgery: mL | Up to 30 weeks after surgery
  Total amount of drainage until drain tube removal Drain tube removal timing: When drainage volume is under 50mL/day for at least 2 days

SECONDARY OUTCOMES:
Total exact drainage volume | Up to 30 weeks after surgery
  total amount volume of drainage bag and amount of aspiration from seroma after drain tube removal
Drainage volume In hospital: mL | Up to 30 weeks after surgery
  Drainage volume In hospital: mL
Total operation running time | Up to 30 weeks after surgery
  Total operation running time
Complication ratio within a month after surgery | Up to 1 year after surgery
  possible pre-defined complications were defined in reference to previous studies
Frequency of seroma aspiration | Up to 30 weeks after surgery
  examination for frequency and total amount of seroma aspiration within a month after surgery. Under 10mL/day, aspiration is stopped

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Seok Park, MD, Study Chair — Yonsei University College of Medicine, Korea
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Bemmel AJ, van de Velde CJ, Schmitz RF, Liefers GJ. Prevention of seroma formation after axillary dissection in breast cancer: a systematic review. Eur J Surg Oncol. 2011 Oct;37(10):829-35. doi: 10.1016/j.ejso.2011.04.012. Epub 2011 Aug 17. PMID 21849243
- [Background] Manouras A, Markogiannakis H, Genetzakis M, Filippakis GM, Lagoudianakis EE, Kafiri G, Filis K, Zografos GC. Modified radical mastectomy with axillary dissection using the electrothermal bipolar vessel sealing system. Arch Surg. 2008 Jun;143(6):575-80; discussion 581. doi: 10.1001/archsurg.143.6.575. PMID 18559751
- [Background] Nespoli L, Antolini L, Stucchi C, Nespoli A, Valsecchi MG, Gianotti L. Axillary lymphadenectomy for breast cancer. A randomized controlled trial comparing a bipolar vessel sealing system to the conventional technique. Breast. 2012 Dec;21(6):739-45. doi: 10.1016/j.breast.2012.08.003. Epub 2012 Sep 7. PMID 22959311
- [Background] Cortadellas T, Cordoba O, Espinosa-Bravo M, Mendoza-Santin C, Rodriguez-Fernandez J, Esgueva A, Alvarez-Vinuesa M, Rubio IT, Xercavins J. Electrothermal bipolar vessel sealing system in axillary dissection: a prospective randomized clinical study. Int J Surg. 2011;9(8):636-40. doi: 10.1016/j.ijsu.2011.08.002. Epub 2011 Sep 10. PMID 21925293
- [Background] Miyagi K, Rossi SH, Malata CM, Forouhi P. Novel use of LigaSure Impact electrosurgical bipolar vessel sealing system in skin-sparing mastectomy. J Plast Reconstr Aesthet Surg. 2015 Jun;68(6):e126-8. doi: 10.1016/j.bjps.2015.01.005. Epub 2015 Jan 26. No abstract available. PMID 25682592
- [Result] Park HS, Lee J, Kim JY, Park JM, Kwon Y. A Prospective Randomized Study to Compare Postoperative Drainage After Mastectomy Using Electrosurgical Bipolar Systems and Conventional Electro-Cautery. J Breast Cancer. 2022 Aug;25(4):307-317. doi: 10.4048/jbc.2022.25.e29. Epub 2022 Jun 27. PMID 35914746